CLINICAL TRIAL: NCT05218460
Title: Evaluation of Methodological and Technical DEvelopmeNts to Improve the Quality and Comfort of Magnetic Resonance Imaging Exam on Voluntary Subjects
Acronym: EDEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Damien MANDRY, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A00243-38
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects will have an MRI examination (Experimental)
  Interventions: Device: MRI examination

INTERVENTIONS:
Device: MRI examination — All subjects (healthy and pathological subjects) will have an MRI examination with a component of the MRI system under development.

SUMMARY:
The EDEN study will make it possible to evaluate one or more development phases (from design to validation through optimization) of a method or a technique on voluntary subjects, in normal or pathological condition.

ELIGIBILITY:
Inclusion Criteria for all subjects :

* to be over 18 year-old,
* to be enrolled in a social security plan,
* to have underwent a pre-inclusion medical examination,
* to give a written consent.

Inclusion Criteria for volunteers with pathology :

- person with a pathology characterized by a functional and / or morphological alteration that may have an impact on the data collected (images, physiological signals, ...).

Exclusion Criteria for all subjects :

* any contraindication to MR examination (active medical device, ferromagnetic foreign body, pregnancy, morbid obesity, claustrophobia, … ),
* subject under a measure of legal protection,
* Person who refuses to be informed by a doctor in th event of a fortuitus discovery of an abnormality on the MRI examination requiring additionnal examinations or specific treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Image quality based on standard imaging quality criteria | 6 months after the last inclusion
  The image quality will be appreciated visually at least by a radiologist or a researcher.
Signal quality based on standard signal quality criteria | 6 months after the last inclusion
  The signal quality will be appreciated visually at least by a radiologist or a researcher.

SECONDARY OUTCOMES:
Comparison of the Signal to Noise Ratio obtained by the component of the MRI system under development and the reference situation. | 6 months after the last inclusion
  ignal to Noise Ratio will be measured in arbitrary units.
Comparison of the Contrast to Noise Ratio obtained by the component of the MRI system under development and the reference situation. | 6 months after the last inclusion
  Contrast to Noise Ratio will be measured in arbitrary units.
Comparison of blurring and artefacts obtained by the component of the MRI system under development and the reference situation. | 6 months after the last inclusion
  Absence of blurring and artefacts will be assessed by at least one radiologist according to an ordinal scale (1 to 5 ; 1 is the worst score and 5 is the better score).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

REFERENCES:
- [Derived] Leclere J, Isaieva K, Drouot G, Gillet R, Felblinger J, Vuissoz PA, Dubernard X. Quantifying symmetry in mandibular condyle motion: a real-time MRI approach. J Oral Facial Pain Headache. 2025 Dec;39(4):227-234. doi: 10.22514/jofph.2025.079. Epub 2025 Dec 12. PMID 41436119